CLINICAL TRIAL: NCT05632172
Title: Influence of Buccal and Palatal Bone Thickness on Post-surgical Marginal Bone Changes Around Implants Placed in Posterior Maxilla
Brief Title: Buccal and Palatal Bone Thickness and Marginal Bone Changes Implants
Acronym: IBPTHPIBC
Status: Completed | Type: Observational
Sponsor: International Piezosurgery Academy (Other)
Collaborators: University of Trieste (Other); University of Messina (Other); University of Campania Luigi Vanvitelli (Other)
Responsible Party: Sponsor
Other Study IDs: maxillary contraction
Record Dates: First submitted 2022-11-20; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Bone Implant; Complications
Keywords: implant; peri-implant bone remodeling; posterior maxilla; bone thickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- maxillary group: implant insertion
  Interventions: Procedure: implant insertion

INTERVENTIONS:
Procedure: implant insertion — bone level dental implant insertion

SUMMARY:
The primary outcome of the study was the vertical variation of peri-implant buccal and palatal bone level from implant placement (T0) to uncovering stage (3 months later - T1)

DETAILED DESCRIPTION:
despite various recommendations, there is insufficient evidence to set a threshold for minimal buccal bone thickness necessary to ensure peri-implant marginal bone stability and optimal aesthetic outcomes.

Therefore, the aim of the present multi-centre prospective study was to investigate the influence of buccal and palatal bone thickness at the time of implant placement on peri-implant bone remodeling during the submerged healing period, with a strict control of possible confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years;
* no smokers;
* no history of periodontal disease;
* healed bone crest (at least six months after tooth extraction);
* crestal bone height ≥8 mm;
* crestal bone with a minimum bucco-palatal width of 6 mm with no concomitant or previous bone augmentation procedures.

Exclusion Criteria:

* absolute contraindications to implant surgery
* immunological or genetic disorders;
* uncontrolled diabetes (HBA1c > 7.5%);
* present or past treatment with anti resorptive drugs;
* oncologic patients;
* history of head or neck radiotherapy;
* alcohol or drugs abuse;
* final insertion torque > 50 Ncm.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patient presenting a single edentulism in the upper premolar area and requiring implant-prosthetic rehabilitation was eligible for this study. Furthermore, patients have to comply with the following inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
peri-implant bone changes in width buccal | three months after surgery
  measurement after implant site preparation with a caliper
peri-implant bone changes in width palatal | three months after surgery
  measurement after implant site preparation with a caliper
peri-implant bone changes in height buccal | three months after surgery
  measurement after implant insertion with a probe
peri-implant bone changes in height palatal | three months after surgery
  measurement after implant insertion with a probe

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Stacchi, Dr, Study Chair — Piezoelectric Surgery Academy
Locations (2):
- Italy (2):
  - Hesire, Cassano Allo Ionio, CS
  - Studio B, Verona, VR

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Merheb J, Quirynen M, Teughels W. Critical buccal bone dimensions along implants. Periodontol 2000. 2014 Oct;66(1):97-105. doi: 10.1111/prd.12042. PMID 25123763
- [Derived] Cicciu M, Pratella U, Fiorillo L, Bernardello F, Perillo F, Rapani A, Stacchi C, Lombardi T. Influence of buccal and palatal bone thickness on post-surgical marginal bone changes around implants placed in posterior maxilla: a multi-centre prospective study. BMC Oral Health. 2023 May 22;23(1):309. doi: 10.1186/s12903-023-02991-3. PMID 37217911